CLINICAL TRIAL: NCT00583856
Title: Is Computer Modeling and Intra-Operative Navigation Helpful With Reconstruction of the Maxillofacial Skeleton?
Brief Title: Computer Modeling With Reconstruction of Maxillofacial Skeleton
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Edward B. Strong, MD, University of California Davis
Other Study IDs: 200614968-1
Record Dates: First submitted 2007-12-22; First posted 2008-01-02 (Estimated); Last update posted 2010-12-20 (Estimated); Status verified 2010-12

CONDITIONS: Maxillofacial Injury
Keywords: computer aided design; maxillofacial fracture; orbital design
MeSH Terms: conditions — Maxillofacial Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Investigator initial study to evaluate the use of preoperative computer modeling and the intraoperative navigation to guide reconstruction of the maxillofacial skeleton.

DETAILED DESCRIPTION:
The concept of open reduction and internal fixation of facial fractures is well accepted. However, there are situations in which an accurate reduction and restoration of facial symmetry is challenging. In these more difficult cases, the PI uses computer aided design/modeling software as well as intra-operative computer aided surgical navigation systems to assist with repair of these complex injuries. A retrospective review of these cases has not previously been performed.

ELIGIBILITY:
Inclusion Criteria:

* specific complex maxillofacial trauma

Exclusion Criteria:

* must meet inclusion criteria

Ages: 11 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: UCDMC Patients with specific complex fractures
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward B Strong, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis, Sacramento, California, United States